CLINICAL TRIAL: NCT05129696
Title: Integrating Early Stimulation and Play at Scale: "MAHAY Mikolo", a Multi-arm Cluster-randomized Controlled Trial
Brief Title: Integrating Early Stimulation and Play at Scale: "MAHAY Mikolo"
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: L'Office National de Nutrition, Madagascar (Unknown); World Bank (Other); University of Nevada, Reno (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-08-12476
Record Dates: First submitted 2021-10-28; First posted 2021-11-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Early Childhood Development
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigators that are analyzing the data are blinded to treatment assignment during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (C): Status quo health and nutrition program (No Intervention)
- Treatment (T): adaption of Reach Up and Learn home visiting program to a group setting (Experimental)
  Interventions: Behavioral: Treatment (T)
- Treatment + (T+): Enhanced play materials/activities package (Experimental)
  Interventions: Behavioral: Treatment + (T+)

INTERVENTIONS:
Behavioral: Treatment (T) — Children area offered to participate in bimonthly group sessions. Each session will have materials and activities appropriate for children spanning a 6-month range (6-12 m, 12-18 m, 12-24 m, 24-30 m) and can accommodate a maximum of 10 children per age group. If more households are interested than can be accommodated by the program, interested families will be randomly selected for participation. A total of 40 children per site will be able to participate in the ECD activities at any one time. With bi-monthly meetings, each child will be exposed to 12 sessions for each age group, and is eligible to transition to the next.
  Arms: Treatment (T): adaption of Reach Up and Learn home visiting program to a group setting
Behavioral: Treatment + (T+) — Caregivers/children participating to the group ECD sessions will be invited to play within a play space equipped with books, and homemade/purchased age-appropriate toys. This will be phased in after 6 months of implementation.
  Arms: Treatment + (T+): Enhanced play materials/activities package

SUMMARY:
The overall objective of the study is to examine the effects of integrating early child development group sessions into the existing, at-scale, community health and nutrition programs administered by the government in Madagascar.

DETAILED DESCRIPTION:
This research is a cluster-randomized trial that will assess the effects of integrating early child development activities on community health worker time use and caregiver time use and participation in the program. The evaluation will compare the addition of early child development sessions to the status quo health and nutrition program, with an additional intervention arm looking at the addition of toys to the program.

This study has four objectives, which will be measured at the community health worker level, and at the caregiver level for caregiver-child dyads (where children are between 6-30 months old at time of intervention launch):

1. Measure how the integration of ECD activities with standard nutrition programming affects the time and task allocation of the community health workers
2. Measure the extent, if any, that the addition of ECD activities crowds out community health worker health/nutrition tasks that are part of the standard community program
3. Measure how the integration of ECD activities affects rates of caregiver participation in nutrition and health activities over time (e.g., during changes in seasonal activities).
4. Measure the impact of enhanced availability and maintenance of age-appropriate play materials/activities on sustained caregiver participation rates in the program.

ELIGIBILITY:
Inclusion Criteria for communities:

1. No other ECD programs present in the community or neighboring communities;
2. At least 40 children monitored at the nutrition center in the target age range of 6-30 months (monitored is defined as attending at least one growth monitoring session between July 2019 to August 2020);
3. Stable supervisory presence. Local NGOs are contracted to monitor and supervise all community health workers and help to strengthen linkages with local structures such as the community health committees and primary care facilities. Each NGO supervisor is in charge to up to 9 communities, which they visit twice a month. The investigators defined stable presence as not having had NGO turnover within the last year.

Among the communities included, children 6-30 months were eligible to participate in the intervention. There was no inclusion criteria for community health workers.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8150 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Community health worker time use | Up to 12 months
  Proportion of working day spent on community health worker activities, measured through recall of hourly time use using monthly phone surveys
Caregiver-child attendance in health and nutrition sessions | Up to 12 months
  Monthly attendance in health and nutrition sessions, measured through session attendance records (0 = Did Not Attend, 1 = Attended)
Caregiver-child attendance in ECD group sessions | Up to 12 months
  Monthly attendance in ECD sessions, measured through session attendance records (0 = Did Not Attend, 1 = Attended)

SECONDARY OUTCOMES:
Community health worker stress | Up to 12 months
  Perceived Stress Scale 4 (PSS-4) administered monthly (Low: 0, High: 16, Higher scores are correlated to more stress)
Community health worker depressive symptoms | Up to 12 months
  Center for Epidemiologic Studies Depression Scale-10 (CESD-10), administered quarterly (Low: 0, High: 30, Higher scores indicate worse symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Galasso, PhD, Principal Investigator — World Bank Group; Lia Fernald, PhD, Principal Investigator — UC Berkeley
Locations (1):
- L'Office National de Nutrition (ONN), Antananarivo, Madagascar

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the World Bank's Open Data and Knowledge Initiative, the deidentified data collected in the study will be made publicly available at the data repository at the World Bank, which is expected to be within 24 months of the final data collection date. Metadata and critical documents (i.e. protocols and questionnaires) will conform to the standards of the Data Documentation Initiative and will be made available within one year of the end of data collection.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Hemlock C, Galasso E, Weber AM, Randriamiarisoa TC, Col M, Dieci M, Ratsifandrihamanana L, Fernald LCH. Integrating early child development into an existing health and nutrition program: evidence from a cluster-randomized controlled trial. BMC Public Health. 2024 Sep 27;24(1):2583. doi: 10.1186/s12889-024-20149-w. PMID 39334156
- [Derived] Galasso E, Ratsifandrihamanana L, Weber AM, Hemlock C, Col M, Dieci M, Rakotomalala N, Rambeloson V, Fernald LCH. Integrating early stimulation and play at scale: study protocol for "MAHAY Mikolo", a multi-arm cluster-randomized controlled trial. BMC Public Health. 2022 Feb 9;22(1):265. doi: 10.1186/s12889-022-12640-z. PMID 35139822